CLINICAL TRIAL: NCT06888921
Title: An Adaptive Clinical Platform Trial to Evaluate the Safety and Efficacy of COM701 as Monotherapy or Combination Therapy as Maintenance Therapy in Participants With Relapsed Platinum Sensitive Ovarian Cancer (PSOC)
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of COM701 in Relapsed Platinum Sensitive Ovarian Cancer
Acronym: MAIA-ovarian
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Compugen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPG-01-201
Record Dates: First submitted 2025-03-12; First posted 2025-03-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Ovarian Cancer Recurrent
Keywords: maintenance therapy; relapsed platinum sensitive ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is an adaptive platform trial enabling the evaluation of COM701 initially as a single agent compared to placebo in relapsed PSOC. This will enable the evaluation of the effects of COM701 as a single agent followed by the potential to adjust the trial to evaluate combinations with COM701.
  A data monitoring committee will review all safety and efficacy data on a regular basis and will make recommendations regarding study unblinding and timing to start additional sub-studies evaluating COM701 in combination with other anti-cancer drugs.
  An interim analysis will be conducted when approximately 60 participants in sub-study 1 have been followed for approximately 9 months.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COM701 (Experimental)
  Interventions: Drug: COM701
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: COM701 — COM701 will be administered via intravenous (IV) infusion once every 3 weeks.
  Arms: COM701
Drug: Normal Saline — Saline will be administered via intravenous (IV) infusion once every 3 weeks
  Arms: Normal Saline

SUMMARY:
The goal of this clinical trial is to learn if the experimental antibody COM701 delays the progression of ovarian cancer in participants with Relapsed Platinum Sensitive Ovarian Cancer. It will also learn about the safety of COM701.

The main questions the trial aims to answer are:

* Does COM701, when used as a maintenance treatment, stop or slow the progression of ovarian cancer?
* Does COM701 delay the time to needing a new anti-cancer treatment?
* What side effects do participants have when taking COM701?

Participants will:

* Visit the clinic once every 3 weeks during which the study treatment will be administered intravenously
* Undergo various tests and procedures to monitor general health throughout the trial including physical examinations, vital sign measurements (heart rate, blood pressure, breathing, and body temperature), weight measurements, electrocardiography (ECG), blood and urine tests and pregnancy tests if relevant.
* Undergo various tests and procedures to assess disease response throughout the trial including tumor imaging by CT scans or MRI to assess the tumor, its location, and size, and the testing of a sample of tumor tissue (from a prior biopsy or a fresh biopsy if feasible, to evaluate tumor response to treatment and to measure levels of tumor markers,

DETAILED DESCRIPTION:
Trial CPG-01-201 is an adaptive-platform trial comprised of multiple sub-studies.

Sub-study 1 will be a parallel group, double-blind, randomized placebo-controlled trial in which participants will be randomized in a 1:2 ratio to either placebo (a look-alike substance that contains no drug) or COM701 treatment arms. This means that there is a 33% chance of being placed in the group getting placebo and a 67% chance of being placed in the group that will get the experimental COM701 antibody.

Subsequent sub-studies will evaluate COM701 in combination with other anti-cancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Has relapsed platinum sensitive epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer
* Has completed at least 2 previous courses (i.e. lines) of platinum-containing therapy
* For the last chemotherapy course prior to being randomized into the study, must have had a minimum of 4 cycles of a platinum containing regimen and achieved a partial or complete tumor response.
* Has received prior maintenance therapy with bevacizumab or a PARP inhibitor if eligible and is not a candidate for, or has declined in writing, bevacizumab or PARP inhibitor therapy.
* Have recovered from toxicities of prior chemotherapy or other therapy (to grade 1 or less, except for alopecia and neuropathy recovered to a ≤grade 2).

Exclusion Criteria:

* Has had 4 or more lines of cytotoxic chemotherapy in total
* Is being treated with immunosuppressive doses of systemic medications, such as steroids within 2 weeks before study drug administration
* Has had prior treatment with PD-1, PD-L1, anti-PVRIG, TIGIT or any other check point inhibitors
* Presence of radiographic or biopsy proven liver metastases at the beginning or completion of current line of platinum-based chemotherapy.
* Drainage of ascites during last 2 cycles of last chemotherapy or any time after completion of the last chemotherapy regimen.
* Bowel obstruction in the 6 weeks prior to randomization.
* Have known active central nervous system metastases and/or carcinomatous meningitis / leptomeningeal carcinomatosis.
* Has active hepatitis B virus (HBV) or hepatitis C virus (HCV), or subjects with human immunodeficiency virus (HIV).
* Has active and clinically relevant bacterial, fungal, or viral infection that is not controlled or requires systemic antibiotics, antifungals, or antivirals, respectively.
* Has received a live viral vaccine within 30 days of planned start of study treatment or requiring a live vaccine during the study.
* Has a history of severe allergic, anaphylactic, or other hypersensitivity reactions to a human or humanized monoclonal antibody (mAb) or allergy to any excipients in the investigational products.
* Has any serious or unstable concomitant systemic disorder
* Has any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the opinion of the investigator, would make the subject inappropriate for entry into the study.
* Is currently participating in or have participated in a clinical study and received an investigational agent or used an investigational device within 4 weeks prior to the first dose of study treatment.
* Is pregnant or breastfeeding or planning to become pregnant during the period of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of COM701 as a single agent on progression free survival when administered as a maintenance regimen in participants with relapsed PSOC | From the date of randomization until the date of disease progression, or date of death from any cause whichever occurs first, assessed up to 2 years
  Progression free survival in COM701-treated participants compared to placebo-treated participants

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the COM701 as a single agent when administered as a maintenance regimen in participants with relapsed PSOC | From randomization up to 90 days post last cycle of study treatment (each cycle is 3 weeks; study treatment may continue up to 2 years).
  Number of participants with adverse events in the COM701 treatment arm compared to the placebo treatment arm
To evaluate the effect of COM701 as a single agent on other efficacy endpoints when administered as a maintenance regimen in participants with relapsed PSOC | From date of randomization until the date of the initiation of a new anti-cancer treatment, or date of death from any cause whichever occurs first, assessed up to 2 years.
  Time to the initiation of a new anti-cancer treatment in COM701-treated participants compared to placebo-treated participants

CONTACTS AND LOCATIONS:
Locations (25):
- United States (11):
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Northwestern Memorial Hospital, Warrenville, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center- Main Campus, New York, New York
  - Ohio State University Wexner Medical Center Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - West Cancer Center, Germantown, Tennessee
  - UVA Comprehensive Cancer Center, Charlottesville, Virginia
- France (8):
  - Centre Hospitalier Regional et Universitaire de Besancon - Hopital Jean-Minjoz, Besançon, France
  - Oncopole Claudius Regaud, Toulouse, France
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Hospices Civils de Lyon- Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de l'Ouest- Site Rene Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
- Israel (6):
  - Assuta Medical Center, Ashdod
  - Rambam Health Care Campus, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah, University Hospital Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Within 12 months of final database lock
Access Criteria: To be decided